CLINICAL TRIAL: NCT04658667
Title: Randomized, Double Blind Evaluation of Late Boost Strategies With IHV01 (FLSC in Aluminum Phosphate) and A244 With or Without ALFQ for HIV-uninfected Participants in the HIV Vaccine Trial RV306 / WRAIR 1920
Brief Title: HIV Vaccine in HIV-uninfected Adults
Acronym: RV546
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Duke University (Other); University of Maryland, Baltimore (Other); Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: S-19-01; RV 546 (Other: MHRP); WRAIR 1920 (Other: USAMRDC/WRAIR)
Record Dates: First submitted 2020-11-23; First posted 2020-12-08 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: HIV
Keywords: HIV Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Full dose IHV01 and A244 (Experimental): Participants will receive a full dose of IHV01 (approximately 300μg) and A244 (approximately 300μg).
  Interventions: Biological: IHV01; Biological: A244
- Fractional dose IHV01 and A244 (Experimental): Participants will receive a fractional dose of IHV01 (approximately 60μg) and A244 (approximately 60μg).
  Interventions: Biological: IHV01; Biological: A244
- Full dose IHV01 and A244 + ALFQ (Experimental): Participants will receive a full dose of IHV01 (approximately 300μg) and A244 (approximately 300μg) plus ALFQ (approximately 0.5mL).
  Interventions: Biological: IHV01; Biological: A244; Biological: ALFQ
- Fractional dose IHV01 and A244 + ALFQ (Experimental): Participants will receive a fractional dose of IHV01 (approximately 60μg) and A244 (approximately 60μg) plus ALFQ (approximately 0.5mL).
  Interventions: Biological: IHV01; Biological: A244; Biological: ALFQ
- Placebo (Placebo Comparator): Normal saline will serve as a placebo for the trial. All placebo injection volumes will match the study vaccine injection volumes for the group in which a participant has been randomized.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IHV01 — IHV01 consists of the Full-Length Single Chain (FLSC) gp120-CD4 chimera subunit HIV-1 vaccine formulated in aluminum phosphate adjuvant. It is encoded by a synthetic gene, which contains a human codon-optimized HIV (BaL) gp120 sequence followed by human CD4D1D2, with a flexible 20-amino acid linker.
  Arms: Fractional dose IHV01 and A244; Fractional dose IHV01 and A244 + ALFQ; Full dose IHV01 and A244; Full dose IHV01 and A244 + ALFQ
Biological: A244 — A244 consists of the gp120 envelope glycoprotein HIV-1 subtype CRF_01AE A244 derived from the CM244 CRF_01AE. The A244 gp120 envelope has an 11 amino N-terminal deletion, similar to the A244 protein used in AIDSVAX B/E. The aluminum hydroxide fluid gel (AHFG) adjuvant that is mixed with A244 consists of Rehydragel HPA that is diluted with sterile water for injection to a concentration of 5 + /- 1mg/mL.
  Arms: Fractional dose IHV01 and A244; Fractional dose IHV01 and A244 + ALFQ; Full dose IHV01 and A244; Full dose IHV01 and A244 + ALFQ
Biological: ALFQ — ALFQ (Army Liposomal Formulation) is a liposomal adjuvant containing a synthetic monophosphoryl lipid A (MPLA) with the addition of QS-21.
  Arms: Fractional dose IHV01 and A244 + ALFQ; Full dose IHV01 and A244 + ALFQ
Other: Placebo — Normal saline (Sodium Chloride for injection USP, 0.9%) will be used as placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether delayed boosting (an extra administration of a vaccine) with the IHV01 (FLSC) protein and A244/AHFG with or without ALFQ will cause the body to make higher amounts of antibodies or different types of antibodies after the vaccination.

DETAILED DESCRIPTION:
The purpose of this study is to define the safety and immunogenicity of IHV01 and A244/AHFG with and without ALFQ at a full dose and at a fractional dose (one-fifth of a full dose) in a late boost setting for participants who had previously received a late boost of AIDSVAX®B/E with or without ALVAC in RV306. Safety will be assessed through the frequency of the overall and specific post-vaccination reactions. Blood, lymph nodes, sigmoid tissue, and mucosal specimens/secretions will be collected to assess humoral, cell-mediated, innate, and mucosal immune responses.

Healthy, HIV-uninfected participants, at a low risk for HIV infection, available for 12 months, who were randomized to receive active vaccine in RV306 and completed all vaccinations will be enrolled. A total of 120 participants will be enrolled across four vaccination groups. In each group, 25 participants will receive IHV01 and A244/AHFG at a full or fractional dose with or without ALFQ and 5 participants will receive placebo. Participants will receive 2 intramuscular (IM) injections into the quadriceps muscle at Day 0. The same quadriceps muscle will be used for both injections. Participants randomized to receive the vaccines will have one injection of IHV01 and one injection of A244/AHFG at a full or fractional dose with or without ALFQ, whereas participants randomized to receive placebo will get 2 separate injections of Normal Saline. All placebo injection volumes will match the vaccine injection volumes for the group in which a participant has been randomized. Participants will be followed-up for up to 12 months after enrollment. Mucosal secretion collections and endocervical cytobrush/swab procedures will be performed at Days 0, 14, 168, and 336 on consenting participants. Leukapheresis, sigmoid biopsy, and lymph node biopsy procedures will be performed only at Day 14 on consenting participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, HIV-uninfected male and female participants
* Prior RV306 recipients who were randomized to receive active vaccine with late boosting at month 12, 15, or 18 and who completed all vaccinations
* Have a Thai identity card
* Must be at low risk for HIV infection per investigator assessment
* Must be able to understand and complete the informed consent process
* Must be capable of reading Thai
* Must successfully complete a Test of Understanding prior to enrollment
* Must be in good general health without clinically significant medical history
* HIV-uninfected per diagnostic algorithm within 45 days of enrollment
* Laboratory screening analysis:

  1. Hemoglobin: Women ≥11.0 g/dL, Men ≥11.5 g/dL
  2. White cell count: 4,000 to 11,000 cells/mm3
  3. Platelets: 150,000 to 450,000/mm3
  4. ALT and AST ≤1.25 institutional upper limit of reference range
  5. Creatinine: ≤1.25 institutional upper limit of reference range
  6. Urinalysis blood and protein no greater than 1+ and negative glucose
* Female-Specific Criteria:

  1. Not currently pregnant or breastfeeding and not planning to become pregnant during the first 3 months after study vaccine/placebo injections
  2. Negative pregnancy test for women at screening, prior to vaccination (same day), and prior to any of the invasive procedures
  3. Be using an adequate birth control method for 45 days prior to receipt of vaccine/placebo and for at least 3 months after receipt of the vaccine/placebo. Adequate birth control is defined as follows: Contraceptive medications delivered orally, intramuscularly, vaginally, or implanted, underneath the skin, surgical methods (hysterectomy or bilateral tubal ligation), condoms, diaphragms, intrauterine device, or abstinence
* Male-Specific Criteria:

  1. Be using an adequate birth control method for at least 3 months after receipt of the vaccine/placebo. For non-vasectomized male participants with female partners of child-bearing potential this includes the use of condoms or abstinence and/or their partner's use of contraceptive medications delivered orally, intramuscularly, vaginally, or implanted, underneath the skin, surgical methods (hysterectomy or bilateral tubal ligation), diaphragms, or intrauterine device.

Exclusion Criteria:

* Asplenia: any condition resulting in the absence of a functional spleen
* Bleeding disorder diagnosed by a medical doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* History of allergic reaction, anaphylaxis, or other serious adverse reaction to vaccines or components of the vaccines
* Volunteer has received any of the following substances:

  1. Chronic use of therapies that may modify immune response, such as IV immune globulin and systemic corticosteroids (in doses of > 20 mg/day prednisone equivalent for periods exceeding 10 days) Note: The following exceptions are permitted and will not exclude study participation: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis; or a short course (duration of 10 days or less, or a single injection) of corticosteroid for a non-chronic condition (based on investigator clinical judgment) at least 14 days prior to enrollment in this study
  2. Blood products within 120 days prior to HIV screening
  3. Immunoglobulins within 30 days prior to HIV screening
  4. Any licensed vaccine within 14 days prior to study vaccine administration in the present study
  5. Receipt of any investigational HIV vaccine other than RV306 products
  6. Investigational research agents or vaccine within 30 days prior to enrollment in the present study
  7. Receipt of a Coronavirus disease 2019 (COVID-19) vaccine that has been given Emergency Use Authorization (or those that become licensed) by the Thai FDA within 14 days prior to study vaccine administration in the present study Note: Volunteers receiving a COVID-19 vaccine that requires 2 doses will not be enrolled until 14 days after the second dose has been administered
  8. Anti-tuberculosis prophylaxis or therapy during the past 90 days prior to enrollment
* Active sexually transmitted infection confirmed by clinical exam and diagnostic test
* Any medical, psychiatric, social condition, occupational reason, or other responsibility that, in the judgment of the investigator, is a contradiction to protocol compliance or impairs a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within 5 years prior to enrollment, a history of suicide ideation or attempt
* Study site employees who are involved in the protocol and/or may have direct access to study related area

Determination of a participants eligibility will be completed at screening. Final evaluation of eligibility will be based on the medical judgment of the principal investigator or designee based on his/her medical and research experience.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Local and Systemic Reactions | Days 0 to 7 post vaccination
  Post-vaccination reactions including erythema, induration, pain/tenderness, swelling and limitation of leg movement, fever, tiredness, chills, myalgia, arthralgia, headache, nausea, and rash will be assessed and recorded on diary cards on Days 0 through 7.
Incidence of Adverse Events, Serious Adverse Events, and Adverse Events of Special Interest (AESIs) as assessed by DAIDS | Days 0 to 336
  Number of participants with Adverse Events on Day 0 through Day 336 as Assessed by Division of AIDS (DAIDS) grading scale and possible attribution to Investigational Product.

SECONDARY OUTCOMES:
Number of Participants with HIV-specific Binding Antibodies | Days 0, 14, 168, and 336.
  Vaccine-induced humoral immune responses are assessed using enzyme-linked immunosorbent assay (ELISA) to detect serum or plasma IgG and IgA binding antibodies to HIV at Days 0, 14, 168, and 336.Humoral mucosal immune responses in the rectal, semen and cervico-vaginal compartments will be assessed using non-invasive sampling methods (sponge, menstrual disc, and masturbation) at the same time points. Cell-mediated immune responses will be assessed utilizing invasive sigmoid and lymph node biopsies that will be performed at Day 14.
Number of Participants with HIV-specific Antigens | Weeks 0, 2, 24, and 48
  Vaccine-induced immune responses are assessed using intracellular cytokine staining (ICS) assays to determine antigen-specific T-cell responses by IFN-gamma and IL-2 at Baseline and weeks 2, 24, and 48.

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, MD, Principal Investigator — Mahidol University; Sorachai Nitayaphan, MD, Principal Investigator — Armed Forces Research Institute of Medical Sciences, Thailand
Locations (2):
- Thailand (2):
  - Armed Forces Research Institute of Medical Sciences, Bangkok
  - Mahidol University, Bangkok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pitisuttithum P, Nitayaphan S, Chariyalertsak S, Kaewkungwal J, Dawson P, Dhitavat J, Phonrat B, Akapirat S, Karasavvas N, Wieczorek L, Polonis V, Eller MA, Pegu P, Kim D, Schuetz A, Jongrakthaitae S, Zhou Y, Sinangil F, Phogat S, Diazgranados CA, Tartaglia J, Heger E, Smith K, Michael NL, Excler JL, Robb ML, Kim JH, O'Connell RJ, Vasan S; RV306 study group. Late boosting of the RV144 regimen with AIDSVAX B/E and ALVAC-HIV in HIV-uninfected Thai volunteers: a double-blind, randomised controlled trial. Lancet HIV. 2020 Apr;7(4):e238-e248. doi: 10.1016/S2352-3018(19)30406-0. Epub 2020 Feb 6. PMID 32035516
- [Background] Rerks-Ngarm S, Pitisuttithum P, Excler JL, Nitayaphan S, Kaewkungwal J, Premsri N, Kunasol P, Karasavvas N, Schuetz A, Ngauy V, Sinangil F, Dawson P, deCamp AC, Phogat S, Garunathan S, Tartaglia J, DiazGranados C, Ratto-Kim S, Pegu P, Eller M, Karnasuta C, Montefiori DC, Sawant S, Vandergrift N, Wills S, Tomaras GD, Robb ML, Michael NL, Kim JH, Vasan S, O'Connell RJ; RV305 Study Team. Randomized, Double-Blind Evaluation of Late Boost Strategies for HIV-Uninfected Vaccine Recipients in the RV144 HIV Vaccine Efficacy Trial. J Infect Dis. 2017 Apr 15;215(8):1255-1263. doi: 10.1093/infdis/jix099. PMID 28329190

DOCUMENTS (3):
  • Study Protocol (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT04658667/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT04658667/SAP_001.pdf
  • Informed Consent Form (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT04658667/ICF_002.pdf